CLINICAL TRIAL: NCT02828696
Title: Minimally Invasive Treatment of Worn Dentition With Innovative CAD-CAM Composites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Mainjot Amélie, Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP001
Record Dates: First submitted 2016-06-15; First posted 2016-07-12 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Tooth Wear
Keywords: CAD-CAM composites; Worn dentition; minimally invasive treatment
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No prep (Other): "No prep" treatment of worn dentition with CAD-CAM composite (PICN)
  Interventions: Device: "No prep" treatment of worn dentition with CAD-CAM composite

INTERVENTIONS:
Device: "No prep" treatment of worn dentition with CAD-CAM composite — Realization of minimally invasive prostheses in PICN (CAD-CAM composite)for worn dentition. Tooth tissues are preserved: no preparation is performed and ultra-thin restorations are CAD-CAM milled.

SUMMARY:
This study evaluates the effectiveness of a minimally invasive treatment, consisting of partial polymer-infiltrated-ceramic-network (PICN) restorations, used in case of rehabilitation of advanced and generalized dental wear over a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting advanced and generalized worn dentition
* All the posterior teeth (minus 2) present wear
* All the anterior teeth (tooth n°13 to n°23) need palatal veneers

Exclusion Criteria:

* More than one missing tooth on each mandible
* Patients with crown(s), bridge(s) or implant(s)
* Patients with non-stabilized parodontite
* Smoker
* Patients suffering from :

  1. Parkinson's Disease
  2. Severe osteoarthritis
  3. Spontaneous pain in the temporomandibular joints, shift of the mandible and an opening limit (25 mm)
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of minimally-invasive treatment protocol of worn dentition | 5 years
  Clinical evaluation following FDI criteria
Quality of life evaluation of minimally-invasive treatment protocol of worn dentition | 5 years
  Quality of life questionnaires

SECONDARY OUTCOMES:
Toxicology evaluation of PICN restorations mechanical and biological behaviour | 5 years
  Toxicology ex vivo evaluation
Wear evaluation of PICN restorations mechanical and biological behaviour | 5 years
  Wear ex vivo evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Mainjot, Study Director — University Hospital Center (CHU) of Liège
Locations (1):
- Institute of Dentistry University of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oudkerk J, Herman R, Eldafrawy M, Wulfman C, Ernst M, Vanheusden A, Mainjot A. Intraoral wear of PICN CAD-CAM composite restorations used in severe tooth wear treatment: 5-year results of a prospective clinical study using 3D profilometry. Dent Mater. 2024 Jul;40(7):1056-1063. doi: 10.1016/j.dental.2024.05.015. Epub 2024 May 18. PMID 38762399